CLINICAL TRIAL: NCT05836415
Title: Effectiveness and Durability Long-term Results of Tricuspid Annuloplasty With 3D Shaped Rings.
Status: Completed | Type: Observational
Sponsor: Michele De Bonis (Other)
Responsible Party: Sponsor-Investigator, Michele De Bonis, Chief of Cardiac Surgery of Advanced and Research Therapies, Ospedale San Raffaele
Organization: Ospedale San Raffaele (Other)
Other Study IDs: EDTA3D
Record Dates: First submitted 2023-01-27; First posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Functional Tricuspid Regurgitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Tricuspid valve annuloplasty with 3D ring — A 3D ring is implanted to treat functional tricuspid valve regurgitation

SUMMARY:
Interest in tricuspid valve disease has grown exponentially over the past few years, in response to increased interest in the poor prognosis of patients with functional tricuspid regurgitation (TR). Tricuspid valve repair (TVR) using a prosthetic ring represents the first option in many centers worldwide, due to the low incidence of residual and recurrent TR and improved survival compared to suture techniques. The goal of ring annuloplasty is to restore the normal geometry of the annulus, thereby improving the coaptation of the leaflets and preventing further dilatation of the annulus. Recently, the three-dimensional geometry of the tricuspid valve has been shown and analyzed by means of data obtained from echocardiography, CT scan and magnetic resonance imaging. Normal tricuspid annulus is characterized by a more prominent part in the anteroseptal commissure area near the aortic valve and right ventricular outflow tract and a deeper part in the posteroseptal commissure area near the coronary sinus ostium . Based on these characteristics, new three-dimensional rings have been developed for tricuspid annuloplasty, such as the MC3 (Edwards Lifescience, Irvine, CA) and the Contour 3D (Medtronic, Minneapolis, MN).

There are few studies concerning the short-term results of tricuspid rings implantation and almost none on the long-term, therefore this study aims to analyze the long-term results of TVR by implantation of the two new prosthetic ring models mentioned above.

The aim of this study is the long-term analysis of the results of tricuspid annuloplasty with three-dimensional rings in patients with functional IT.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Operated for functional TR
* Implantation of three-dimensional tricuspid prosthetic ring MC3 or Contour 3D, isolated or concomitant to surgery on the left heart sections
* Surgical access in median sternotomy or minithoracotomy

Exclusion Criteria:

- emergency/urgency intervention

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who underwent tricuspid surgery due to functional tricuspid regurgitation, treated with implant of a 3D ring
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2020-12-29 (Actual); Study Completion 2020-12-29 (Actual)

PRIMARY OUTCOMES:
Mortality | through study completion, an average of 7 years

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No